CLINICAL TRIAL: NCT01875367
Title: Phase III Trial to Evaluate Patient´s Preference of Subcutaneous Trastuzumab vs Intravenous (IV) Administration in HER2 Positive Advanced Breast Cancer Who Have Received IV Trastuzumab at Least 4 Months and Without Disease Progression
Brief Title: Phase III to Evaluate Patient´s Preference of Subcutaneous Trastuzumab vs Intravenous in HER2+ Advanced Breast Cancer
Acronym: ChangHER-SC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2012-07; 2012-004928-38 (EudraCT Number)
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
Keywords: Subcutaneous trastuzumab; Intravenous trastuzumab; HER2 positive; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Intervention Model Description: Eligible patients, from the randomization and before starting subcutaneous trastuzumab (SC-t), received an additional intravenous (IV-t) cycle. After receiving this cycle, patients started the treatment with the study medication, SC-t at a fixed dose of 600 mg every 3 weeks (+3 days) for 4 cycles (2 administered from the injection of a vial in a syringe and 2 with the single-use injection device [SID]), being randomized 1:1 in two arms of treatment without washout period:
  * Arm A (1 cycle of IV-t followed by 2 cycles of SC-t with vial followed by 2 cycles of SC-t with SID)
  * Arm B (1 cycle of IV-t followed by 2 cycles of SC-t with SID followed by 2 cycles of SC-t with vial)
  This is not a cross-over study.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: T-IV + T-SC vial + T-SC device (Experimental): Trastuzumab intravenous (T-IV) x 1 cycle (usual dose of Trastuzumab), followed by 600mg of Trastuzumab Subcutaneous (T-SC) with vial (Injectable Solution) x 2 cycles, followed by 600mg of T-SC with single injection device (SID) x 2 cycles.
  Interventions: Drug: Trastuzumab Injectable Solution; Drug: Trastuzumab Injectable Product; Drug: Trastuzumab Injection
- Arm B: T-IV + T-SC device + T-SC vial (Experimental): Trastuzumab intravenous (T-IV) x 1 cycle (usual dose of Trastuzumab), followed by 600mg of Trastuzumab Subcutaneous (T-SC) with single injection device (SID) x 2 cycles, followed by 600mg of T-SC with vial (Injectable Solution) x 2 cycles.
  Interventions: Drug: Trastuzumab Injectable Solution; Drug: Trastuzumab Injectable Product; Drug: Trastuzumab Injection

INTERVENTIONS:
Drug: Trastuzumab Injectable Solution — Subcutaneous injection vial with a fixed dose of trastuzumab (600mg) and recombinant human hyaluronidase (10.000U) identical to that provided by the device. 3 weeks x 2 cycles.
  Other Names: Herceptin
Drug: Trastuzumab Injectable Product — Single injection device is provided and loaded with the mixture of trastuzumab (600mg) and recombinant human hyaluronidase (10.000U) and is ready for use. 3 weeks x 2 cycles
  Other Names: Herceptin
Drug: Trastuzumab Injection — Powder for concentrate for solution for infusion. 1 cycle
  Other Names: Herceptin

SUMMARY:
GEICAM/2012-07 is a study phase III, prospective, open, randomized, multicenter and national designed to assess patient preference for intravenous (IV) or subcutaneous (SC) of trastuzumab, and within the SC by the administration through the vial or device self-administration in patients with disseminated breast cancer HER2.

DETAILED DESCRIPTION:
Approximately 195 patients will be included to receive subcutaneous trastuzumab a fixed dose of 600 mg every 3 weeks for 4 cycles (2 administered from the injection of a vial with a syringe and 2 with the injection device). Following administration of these four cycles, the patient will decide whether or not to continue with the subcutaneous formulation of trastuzumab every 3 weeks until progression (out of the study). Since the randomization in the study until the start with subcutaneous trastuzumab, patients will receive a treatment cycle of intravenous trastuzumab as usual.

Main objective: Proportion of patients indicate a preference for the use of subcutaneous vs intravenous trastuzumab.

This principal primary objective will be analyzed with the answers to questionnaire of experiences and preferences of the patients (Principal endpoint) The duration of the study has been estimated after 34 months.

ELIGIBILITY:
Inclusion Criteria:

* Woman, 18 years old or upper.
* Patient with advanced breast cancer with human epidermal growth factor receptor 2 (HER 2) positive histologically confirmed. The criteria for positivity HER 2 are:

  1. immuno-histochemistry (IHC) 3+ (>10% of tumor cells with complete and intense membrane staining)
  2. IHC 2+ with fluorescent in situ hybridization (FISH) / Chromogenic in situ hybridization (CISH) / silver-enhanced in situ hybridization (SISH) + for HER 2 amplification (*)
  3. FISH / CISH / SISH + for HER 2 amplification (*) (*) Defined as the ratio of copies of HER 2/neu and copies of centromere of chromosome 17 (CEP17)> 2.2, or a number of copies of HER 2/neu> 6, as per local laboratory criteria.
* Patient receiving trastuzumab with or without chemotherapy or hormonal therapy for at least 4 months.
* No evidence of disease progression (clinical and / or radiological) for at least 4 months before inclusion in the study and with a life expectancy of at least 3 months.
* Adequate performance status: Eastern Cooperative Oncology Group (ECOG) <2.
* Adequate bone marrow function, liver and kidney
* Proper cardiac function (LVEF within normal limits the center, measured by echocardiography or MUGA).
* The patient must have been informed of the study and must sign and date informed consent document for entry into the trial.
* The patient must be willing and able to comply with study procedures and be available to answer the study questionnaires.

Exclusion Criteria:

* Patients with no advanced breast cancer.
* Breast cancer patients with tumors HER 2-negative.
* The patient has another active malignancy other than breast adenocarcinoma; are excluded the non-melanoma skin cancer or any other properly treated in situ neoplasia. Patients with a history of malignancy, if they bear> 5 years without evidence of disease could be included.
* The patient has uncontrolled brain metastases.
* Concomitant administration, or in the 4 weeks prior to study entry, of other experimental treatment.
* Known hypersensitivity to trastuzumab or to any of its components.
* Patients with severe dyspnea at rest or requiring supplemental oxygen.
* Heart disease or serious medical pathological prevent trastuzumab administration: documented history of congestive cardiac insufficiency (CCI), high-risk arrhythmias uncontrolled angina requiring medication, clinically significant valvular disease, history of myocardial infarction or evidence of transmural infarction on ECG or hypertension poorly controlled.
* Presence of any concomitant serious systemic disease that is incompatible with the study (at the discretion of the investigator).
* The patient is pregnant or lactating. Women of childbearing potential should undergo pregnancy testing blood or urine within 14 days prior to inclusion as institutional rules and use a non-hormonal contraceptive suitable: intrauterine device, barrier method (condom or diaphragm) also used in conjunction with spermicidal cream, total abstinence or surgical sterilization, during treatment with the study drugs and for 6 months following the end of treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-09-18 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospitales Universitarios Virgen del Rocío
Locations (27):
- Spain (27):
  - Hospital de Manacor, Manacor, Balearic Islands
  - Hospital General Universitario de Granollers, Granollers, Barcelona
  - Hospital de Mataró, Mataró, Barcelona
  - Hospital Sant Joan Despí Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital Virgen del Puerto de Plasencia, Plasencia, Cáceres
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Univesitario Quirón Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Santa Lucía, Cartagena, Murcia
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital Universitario San Joan de Reus, Reus, Tarragona
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Result] Ciruelos EM, Montano A, Rodriguez CA, Gonzalez-Flores E, Lluch A, Garrigos L, Quiroga V, Anton A, Malon D, Chacon JI, Velasco M, Gonzalez-Cortijo L, Jolis L, Echarri MJ, Munoz M, Pascual T, Amigo Y, Casas M, Carrasco E, Casas A. Phase III study to evaluate patient's preference of subcutaneous versus intravenous trastuzumab in HER2-positive metastatic breast cancer patients: Results from the ChangHER study (GEICAM/2012-07). Eur J Cancer Care (Engl). 2020 Jul;29(4):e13253. doi: 10.1111/ecc.13253. Epub 2020 Jun 23. PMID 32578279
- See also: Sponsor's web — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients, from the randomization and before starting subcutaneous trastuzumab (SC-t), received an additional intravenous (IV-t) cycle. After receiving this cycle, patients started the treatment with the study medication, SC-t at a fixed dose of 600 mg every 3 weeks (+3 days) for 4 cycles (2 administered from the injection of a vial in a syringe and 2 with the single-use injection device [SID]), being randomized 1:1 in two arms of treatment without washout period.
Pre-assignment Details: This is not a cross-over study.
Period: Overall Study
Arm/Group | Arm A: T-IV + T-SC Vial + T-SC Device | Arm B: T-IV + T-SC Device + T-SC Vial
Started | 81 | 85
Completed | 76 | 83
Not Completed | 5 | 2
Not completed — Not complete at least 2 questionaries | 4 | 2
Not completed — Not receive study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: T-IV + T-SC Vial + T-SC Device | Arm B: T-IV + T-SC Device + T-SC Vial | Total
Number analyzed (Participants) | 81 | 85 | 166
Age, Continuous [Median (Full Range); unit: years] | 63 [35 to 93] | 58 [38 to 85] | 60 [35 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 85 | 166
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 78 | 83 | 161
  Black | 1 | 0 | 1
  Hispanic | 1 | 0 | 1
  Arabian | 1 | 2 | 3
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 8 | 12 | 20
  Postmenopausal | 73 | 73 | 146
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — Measure Description: ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death.
  0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 63 | 61 | 124
    ECOG 1 | 17 | 24 | 41
    ECOG 2 | 1 | 0 | 1
Estrogen Receptor [Count of Participants; unit: Participants] — A cancer is called hormonal receptor positive if it has receptors for progesterone or estrogen. This suggests that the cancer cells, like normal breast cells, may receive signals from progesterone or estrogen that could promote their growth.
  If the cancer is hormone-receptor-negative (no receptors are present), then hormonal therapy is unlikely to work.
  Participants
    Positive | 46 | 60 | 106
    Negative | 35 | 25 | 60
Progesterone Receptor [Count of Participants; unit: Participants] — A cancer is called hormonal receptor positive if it has receptors for progesterone or estrogen. This suggests that the cancer cells, like normal breast cells, may receive signals from progesterone or estrogen that could promote their growth.
  If the cancer is hormone-receptor-negative (no receptors are present), then hormonal therapy is unlikely to work.
  Participants
    Negative | 50 | 38 | 88
    Positive | 31 | 47 | 78
Time with IV trastuzumab for metastasis at registration [Median (Full Range); unit: years] | 1.9 [0.35 to 13.67] | 1.78 [0.34 to 14.05] | 1.8 [0.34 to 14.05]
Treatment/s combined with IV-trastuzumab at registration [Count of Participants; unit: Participants]
  Homonotherapy (HT) | 34 | 36 | 70
  Chemotherapy (CT) | 12 | 9 | 21
  Other anti-cancer therapy | 7 | 10 | 17
  Other anti-cancer therapy+CT | 2 | 4 | 6
  Other anti-cancer therapy+HT | 2 | 2 | 4
  None | 24 | 24 | 48
Other anti Human Epidermal growth factor Receptor 2 (HER-2) therapy at registration [Count of Participants; unit: Participants]
  Pertuzumab | 8 | 11 | 19
  Lapatinib | 3 | 5 | 8
  None | 70 | 69 | 139
Administration route at registration [Count of Participants; unit: Participants]
  Intravenous | 25 | 27 | 52
  Intramuscular | 5 | 5 | 10
  Subcutaneous | 4 | 5 | 9
  Oral | 25 | 29 | 54
  None | 22 | 19 | 41
Metastases 1 at diagnosis [Count of Participants; unit: Participants]
  No | 53 | 52 | 105
  Yes | 28 | 33 | 61
Visceral metastases at registration [Count of Participants; unit: Participants]
  Yes | 41 | 49 | 90
  No | 40 | 36 | 76
Bone metastases at registration [Count of Participants; unit: Participants]
  Yes | 34 | 41 | 75
  No | 47 | 44 | 91
Skin/soft tissue/lymph nodes metastases at registration [Count of Participants; unit: Participants]
  Yes | 31 | 29 | 60
  No | 50 | 56 | 106
Median of prior treatment lines at registration [Median (Full Range); unit: Treatment lines] — The greater number of lines previously received by a patient, the worst prognosis.
  Treatment lines | 1 [0 to 7] | 1 [1 to 7] | 1 [0 to 7]
Prior treatment lines at registration [Number; unit: participants] — The greater number of lines previously received by a patient, the worst prognosis.
  participants
    1 Line | 48 | 55 | 103
    2 Lines | 19 | 10 | 29
    3 Lines | 6 | 9 | 15
    4 Lines | 4 | 6 | 10
    5 Lines | 1 | 2 | 3
    6 Lines | 1 | 2 | 3
    7 Lines | 1 | 1 | 2
    None Line | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Subcutaneous vs. Intravenous Treatment Preference
Description: The percentage of patients who indicate a preference for the use of the intravenous vs subcutaneous administration of trastuzumab was analyzed with the answer to the questionnaire C2, question number 39 (All things considered, what method of administration do you prefer? Subcutaneous; Intravenous; No preference) of experiences and preferences of the patient.
Time Frame: Up to 12 weeks
Population: Patients were randomized 1:1 in 2 arms:
  Arm A: (1 cycle IV-t followed by 2 cycles SC-t with vial followed by 2 cycles SC-t with SID) Arm B: (1 cycle IV-t followed by 2 cycles SC-t with SID followed by 2 cycles SC-t with vial)
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: T-IV + T-SC Vial + T-SC Device | Arm B: T-IV + T-SC Device + T-SC Vial
Number analyzed (Participants) | 76 | 83
Participants
  Subcutaneous | 66 | 71
  Intravenous | 6 | 5
  No preference | 4 | 7

2. Secondary Outcome: Percentage of Participants With Subcutaneous Treatment (Vial vs Device Administration) Preference
Description: The percentage of patients who indicate a preference for the use of SC administration by vial or device was analyzed. This was discussed in the answer to questionaire C3, question number 28 (All things considered, what method of administration do you prefer? Subcutaneous; Intravenous; No preference) of the questionnaire of experiences and preferences of the patient.
Time Frame: Up to 12 weeks
Population: Patients were randomized 1:1 in 2 arms:
  Arm A: (1 cycle IV-t followed by 2 cycles SC-t with vial followed by 2 cycles SC-t with SID) Arm B: (1 cycle IV-t followed by 2 cycles SC-t with SID followed by 2 cycles SC-t with vial) It has been analysed in patients from Intention To Treat (ITT) population which have completed questionnaire nº 3 (Arm A 72 patients and Arm B 80 patients).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: T-IV + T-SC Vial + T-SC Device | Arm B: T-IV + T-SC Device + T-SC Vial
Number analyzed (Participants) | 72 | 80
Participants
  Device | 46 | 44
  Vial | 20 | 20
  No preference | 4 | 13
  Not answered | 2 | 3

3. Secondary Outcome: Percentage of Medical Staff With Intravenous vs. Subcutaneous Preference
Description: The medical staff satisfaction was analyzed with the answers to question number 33a (Considering all aspects, with what method of administration were you more satisfied? Between Intravenous vs. Subcutaneous: Intravenous; Subcutaneous; No differences) of the questionnaire of experiences and preferences of the medical staff.
  Health care professionals were not considered enrolled, but did contribute to this assessment.
Time Frame: Up to 12 weeks
Population: Questionnaires were given to the health care professionals of both arms. Information has been analyzed per administration type, not per arm.
  39 health care professional satisfaction questionnaires were completed. Health care professionals were not considered enrolled, but did contribute to this assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Both Arms: Questionnaires were given to the health care professionals of both arms. There have been completed 39 health care professional satisfaction questionnaires. Information not provided by arm.
Arm/Group | Both Arms
Number analyzed (Participants) | 39
Participants
  Subcutaneous | 34
  Intravenous | 0
  No differences | 4
  Not answered | 1

4. Secondary Outcome: Percentage of Medical Staff Subcutaneous Device vs. Vial Preference
Description: The medical staff satisfaction was analyzed with the answers to question number 33b (Considering all aspects, with what method of administration were you more satisfied? Between Vial vs. Device: Preferred device; Preferred vial; No Preference) of the questionnaire of experiences and preferences of the medical staff. Health care professionals were not considered enrolled, but did contribute to this assessment.
Time Frame: Up to 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Both Arms
Number analyzed (Participants) | 39
Participants
  Preferred device | 20
  Preferred vial | 11
  No Preference | 8

5. Secondary Outcome: Patient Time in Healthcare Unit and Sitting in Chair/Bed
Description: Time spent by patient in the healthcare unit: Time between entrance and exit from the healthcare unit.
  Time spent by patient sitting in the infusion/treatment chair/bed: Time between sitting and rising from the patient treatment chair/bed The data was collected by qualified observers from site staff that measured the time spent by healthcare professional using a chronometer, and write it down in the paper questionnaires or directly or after in the electronic case report form.
Time Frame: An average of 4 months
Population: This analysis was considered from 87 patients of the 166 patients included into the study, on who information of observed tasks were collected. 217 observations were made from these patients: 74 about IV-t administration process, 75 about SC-SID administration process, 68 about SC-Vial administration process.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Observations
Groups:
- Both Arms: Intravenous-Trastuzumab (IV-t): Patients from both arms (A and B) who received Intravenous-Trastuzumab as per clinical practice.
- Both Arms: Subcutaneous-Trastuzumab Vial (SC-t Vial): Patients from both arms (A and B) who received Subcutaneous (SC) injection vial.
- Boths Arms: Subcutaneous-Trastuzumab Device (SC-t SID): Patients from both arms (A and B) who received Single injection device
Arm/Group | Both Arms: Intravenous-Trastuzumab (IV-t) | Both Arms: Subcutaneous-Trastuzumab Vial (SC-t Vial) | Boths Arms: Subcutaneous-Trastuzumab Device (SC-t SID)
Number analyzed (Participants) | 87 | 87 | 87
Number analyzed (Observations) | 74 | 75 | 68
minutes
  Healthcare unit | 203 (123.57) | 144.84 (121.99) | 122.9 (112.33)
  Sitting in the infusion/treatment chair/bed | 100.01 (56.34) | 31.6 (28.74) | 24.75 (15.42)

6. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE)
Description: Safety was assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 4.03.
Time Frame: Through study treatment, an average of 12 weeks
Population: Safety Population included all patients randomized in the study who received at least one dose of treatment, and they were analyzed according to the actual treatment received (81 patients in arm A and 85 patients in arm B).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: T-IV + T-SC Vial + T-SC Device | Arm B: T-IV + T-SC Device + T-SC Vial
Number analyzed (Participants) | 81 | 85
Participants | 76 | 84

ADVERSE EVENTS:
Time Frame: Through study treatment, an average of 12 weeks
Description: AE were reported after Informed Consent Document (ICD) and before study drugs until approximately 30 days following the discontinuation of study treatment.
  AEs were recorded for each Arm group Arm A and Arm B, so information can not be provided separately per intervention.
Arm/Group | Arm A: T-IV + T-SC Vial + T-SC Device | Arm B: T-IV + T-SC Device + T-SC Vial
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/85
Serious Adverse Events (participants affected / at risk) | 2/81 | 10/85
Other Adverse Events (participants affected / at risk) | 76/81 | 84/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: T-IV + T-SC Vial + T-SC Device (N=81) | Arm B: T-IV + T-SC Device + T-SC Vial (N=85)
Fever (General disorders) | 1 | 0
Heart failure (Cardiac disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Nodule in left breast (Reproductive system and breast disorders) | 0 | 1
Cold (Infections and infestations) | 0 | 1
Nodule in right breast (Reproductive system and breast disorders) | 0 | 1
Lack of strength in left leg (Musculoskeletal and connective tissue disorders) | 0 | 1
Catheter related infection (Bacteriemia) (Infections and infestations) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Surgery for surgical castration (Reproductive system and breast disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ostenecrosis produced by biphosphonates (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: T-IV + T-SC Vial + T-SC Device (N=81) | Arm B: T-IV + T-SC Device + T-SC Vial (N=85)
Platelet count decreased (Investigations) | 1 | 0 — Grade 4
Platelet count decreased (Investigations) | 4 | 8 — Grade 1
Creatinine increased (Investigations) | 0 | 1 — Grade 4
Creatinine increased (Investigations) | 1 | 2 — Grade 2
Creatinine increased (Investigations) | 13 | 17 — Grade 1
Alanine aminotransferase increased (Investigations) | 0 | 1 — Grade 3
Alanine aminotransferase increased (Investigations) | 0 | 1 — Grade 2
Alanine aminotransferase increased (Investigations) | 16 | 10 — Grade 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 — Grade 3
Aspartate aminotransferase increased (Investigations) | 15 | 17 — Grade 1
Fatigue (General disorders) | 0 | 1 — Grade 3
Fatigue (General disorders) | 3 | 5 — Grade 2
Fatigue (General disorders) | 10 | 16 — Grade 1
Heart failure (Cardiac disorders) | 0 | 1 — Grade 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 — Grade 3
Nodule in left breast (Reproductive system and breast disorders) | 0 | 1 — Grade 3
Alkaline phosphatase increased (Investigations) | 1 | 0 — Grade 3
Alkaline phosphatase increased (Investigations) | 1 | 2 — Grade 2
Alkaline phosphatase increased (Investigations) | 12 | 15 — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 — Grade 3
Diarrhea (Gastrointestinal disorders) | 0 | 4 — Grade 2
Diarrhea (Gastrointestinal disorders) | 6 | 5 — Grade 1
Hemoglobin increased (Investigations) | 1 | 0 — Grade 3
Neutrophil count decreased (Investigations) | 7 | 5 — Grade 2
Neutrophil count decreased (Investigations) | 13 | 13 — Grade 1
Neutrophil count decreased (Investigations) | 2 | 0 — Grade 3
Nausea (Gastrointestinal disorders) | 1 | 0 — Grade 3
Nausea (Gastrointestinal disorders) | 1 | 0 — Grade 2
Nausea (Gastrointestinal disorders) | 4 | 6 — Grade 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Grade 3
Vomiting (Gastrointestinal disorders) | 1 | 0 — Grade 3
Vomiting (Gastrointestinal disorders) | 2 | 0 — Grade 2
Vomiting (Gastrointestinal disorders) | 1 | 0 — Grade 1
White blood cells decreased (Investigations) | 7 | 5 — Grade 2
White blood cells decreased (Investigations) | 15 | 17 — Grade 1
Anemia (Blood and lymphatic system disorders) | 5 | 2 — Grade 2
Anemia (Blood and lymphatic system disorders) | 27 | 32 — Grade 1
Injection site reaction (General disorders) | 2 | 3 — Grade 2
Injection site reaction (General disorders) | 9 | 6 — Grade 1

LIMITATIONS AND CAVEATS:
We do not have longterm follow-up data of the SC-t efficacy. Device SC-t SID has not been commercialized. All patients had already been treated with IV-t for at least 4 months without disease progression prior to the study entry.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less